CLINICAL TRIAL: NCT06075615
Title: A Multicenter, Observational Study to Describe the Effectiveness and Treatment Patterns of Dacomitinib Among Epidermal Growth Factor Receptor Mutation-Positive Non-Small Cell Lung Cancer Patients With Brain Metastasis
Brief Title: A Study to Learn About Dacomitnib in Patients With Non-small Cell Lung Cancer Which Has Spread to the Brain.
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A7471072; NCT06075615 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-09-18; First posted 2023-10-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Dacomitinib, Non-Small Cell Lung Cancer, Brain Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- dacomitnib
  Interventions: Drug: dacomitnib

INTERVENTIONS:
Drug: dacomitnib — patients with dacomitnib as first line treatment for advanced NSCLC with brain metastasis

SUMMARY:
The purpose of this study is to learn about dacomitinib for the possible treatment of lung cancer which has spread to other parts of the body.

This study is seeking participants who:

* have lung cancer that has reached at least the brain.
* have a type of gene called epidermoid growth factor receptor. A gene is a part of your DNA that has instructions for making things your body needs to work.
* have not received any treatment before.

All participants in this study will receive dacomitnib 1 time a day. Dacomitinib is a tablet that is taken by mouth at home. They can continue to take dacomitnib until their cancer is no longer responding. The study will look at the experiences of people receiving the study medicine. This will help to see if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* confirmed diagnosis of EGFR mutation-positive NSCLC
* at least one measurable intracranial metastasis
* ECOG-PS of 0, 1 or 2
* dacomitinib as first-line treatment for advanced NSCLC
* Evidence of a personally signed and dated informed consent document (ICD)

Exclusion Criteria:

* any anti-cancer systemic treatment within 12 months prior to index date
* currently on active investigational drug(s) treatment in other clinical studies (Phase 1-4) within 2 weeks before the current study begins and/or during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with epidermoid growth factor receport (EGFR)-positive non-small cell lung cancer (NSCLC) with brain metastasis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
The real-world intracranial overall response rate (rwICORR) at Month 3 | 3 months from first dose of dcomitnib
  The percentage of patients achieving real-world intracranial overall response (complete response (CR) or partial response (PR)) for brain metastases at Month 3 (± 4 weeks) will be summarized.
The real-world intracranial overall response rate (rwICORR) at Month 6 | 6 months from first dose of dacomitnib
  The percentage of patients achieving real-world intracranial overall response (CR or PR) for brain metastases at Month 6 (± 4 weeks) will be summarized.
The real-world intracranial overall response rate (rwICORR) at Month 12 | 12 months from first dose of dacomitinib
  The percentage of patients achieving real-world intracranial overall response (CR or PR) for brain metastases at Month 12 (± 4 weeks) will be summarized.
The real-world intracranial clinical benefit rate (rwICBR) at Month 3 | 3 months from first dose of dacomitinib
  The percentage of patients with real-world intracranial clinical benefit (CR, PR or SD) for brain metastases at Month 3 (± 4 weeks) will be summarized
The real-world intracranial clinical benefit rate (rwICBR) at Month 6 | 6 months from first dose of dacomitinib
  The percentage of patients with real-world intracranial clinical benefit (CR, PR or SD) for brain metastases at Month 6 (± 4 weeks) will be summarized
The real-world intracranial clinical benefit rate (rwICBR) at Month 12 | 12 months from first dose of dacomitinib
  The percentage of patients with real-world intracranial clinical benefit (CR, PR or SD) for brain metastases at Month 12 (± 4 weeks) will be summarized
The real-world intracranial time to progression (rwICTTP) | 30 months from first dose of dacomitinib
  The mean and median of the time to the date of the first documentation of real-world progression of intracranial disease.
The real-world systemic overall response rate (rwORR) at Month 3 | 3 months from first dose of dacomitinib
  The number and percentage of patients achieving real-world systemic overall response (CR or PR) for brain metastases at Month 3 (± 4 weeks) will be summarized.
The real-world systemic overall response rate (rwORR) at Month 6. | 6 months from first dose of dacomitinib
  The number and percentage of patients achieving real-world systemic overall response (CR or PR) for brain metastases at Month 6 (± 4 weeks) will be summarized.
The real-world systemic overall response rate (rwORR) at Month 12. | 12 months from first dose of dacomitinib
  The number and percentage of patients achieving real-world systemic overall response (CR or PR) for brain metastases at Month 12 (± 4 weeks) will be summarized.
The real-world progression-free survival (rwPFS) during 12 months from index date | 12 months from index date
  Time to real-world disease progression or death, whichever occurs first, during 12 months from index date will be summarized by the K-M plot with the corresponding 95% CI.
The real-world overall survival (rwOS) during 12 months from index date | 12 months from index date
  Time to real-world death during 12 months from index date will be summarized by the K-M plot with the corresponding 95% CI.
The real-world overall survival (rwOS) during 24 months from index date | 24 months from index date
  Time to real-world death during 24 months from index date will be summarized by the K-M plot with the corresponding 95% CI.

SECONDARY OUTCOMES:
Percentage of patients with dacomitinib treatment discontinuation | 30 months from first dose of dacomitinib
  The percentage of patients with dacomitinib treatment discontinuation for any reason during follow-up period will be summarized.
Time to dacomitinib treatment discontinuation | 30 months from first dose of dacomitinib
  Time to dacomitinib treatment discontinuation during follow-up period will be summarized by the K-M plot with the corresponding 95% CI.
Number of patients with dacomitinib dosage change and reasons | 30 months from first dose of dacomitinib
  The number of patients with dacomitinib dosage change and reason during follow-up period will be summarized.
Time to dacomitinib dosage change | 30 months from first dose of dacomitinib
  Time to dacomitinib dosage change during follow-up period will be summarized by the K-M plot with the corresponding 95% CI.
Concomitant NSCLC-related treatment | 30 months from first dose of dacomitinib
  The number patients with concomitant NSCLC-related treatment will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.